CLINICAL TRIAL: NCT00157716
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Multi-Center Study to Evaluate the Cardiovascular and Cerebrovascular Effects of MC-1 in Patients Undergoing High-Risk Coronary Artery Bypass Graft (CABG) Surgery
Brief Title: MEND-CABG (MC-1 to Eliminate Necrosis and Damage in Coronary Artery Bypass Graft Surgery)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicure (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MC6021-CR-03-02
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-10-31 (Estimated); Status verified 2006-10

CONDITIONS: Coronary Artery Bypass Graft Surgery; Myocardial Ischemia; Reperfusion Injury; Myocardial Revascularization
Keywords: Coronary; surgery; ischemia; reperfusion injury; cardiac; heart; neurological; cardiopulmonary bypass; cardioprotection
MeSH Terms: conditions — Myocardial Ischemia; Reperfusion Injury; Ischemia; Neurologic Manifestations | interventions — Pyridoxal Phosphate

INTERVENTIONS:
Drug: (MC-1) Pyridoxal-5'-phosphate

SUMMARY:
The purpose of this study is to determine whether MC-1 is effective and safe in reducing cardiovascular and neurological events in patients undergoing high-risk coronary artery bypass surgery

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) effectively relieves angina, results in longer survival, and a better quality of life in specific subgroups of patients with obstructive coronary artery disease. Due to the high incidence of coronary artery disease worldwide, as well as the effectiveness of the surgical procedure, CABG surgery makes up one of the top ten most frequently performed procedures in North America and Europe. In the United States it is estimated that over 700,000 CABG procedures are performed per year.

Despite the benefits of CABG surgery, patients undergoing these procedures may also suffer serious adverse outcomes including operative mortality, myocardial infarction, unstable angina, ventricular failure, life-threatening arrhythmia, renal insufficiency, and stroke.

Some of the proposed causes of cardiovascular morbidity and mortality after CABG include perioperative ischemia, inadequate myocardial protection and reperfusion injury. The impact of these serious complications is significant. Incidence rates of death and MI following CABG surgery range from 5% to 12% depending on risk status. Results from large clinical trials have recently demonstrated the importance of neurologic deficits as a problematic outcome of CABG. These deficits include memory impairment, psychomotor, visuospatial, attention and language abilities as measured by neuropsychological testing as well as sensori-motor abnormalities associated with stroke.

MC-1 is a naturally occurring small molecule. Evidence from pre-clinical and clinical studies suggests that MC-1 protects the heart from ischemic damage and ischemia-reperfusion injury. This trial will assess the effects of MC-1 compared to placebo on cardiovascular and neurological events following CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients must be scheduled to undergo CABG surgery (during routine scheduling times) planned to use cardiopulmonary bypass

Patients must be considered at high risk for subsequent neurological or myocardial complications defined as meeting 2 or more of the following:

* Age >65
* Current smoker
* History of diabetes mellitus requiring treatment other than diet
* Evidence of left ventricular dysfunction or congestive heart failure assessed by: ejection fraction (EF) <45%, left ventricular end diastolic pressure (LVEDP) or pulmonary wedge pressure greater than or equal to 20 mm Hg, pulmonary edema by chest X-ray, cardiothoracic ratio >50% on chest X-ray
* History of a previous non-disabling stroke, transient ischemic attack, or carotid endarterectomy
* Urgent CABG intervention defined as the need to stay in the hospital (although patient may be operated on within a normal scheduling routine
* History of a myocardial infarction that occurred more than 48 hours but less than 6 weeks prior to CABG surgery
* Prior peripheral artery surgery or angioplasty
* Moderate renal dysfunction defined by creatinine ≥ 133 micromol/L (1.5 mg/dL), but < 250 micromol/L (2.8 mg/dL)
* Presence of at least one asymptomatic carotid artery stenosis (≥50%) either in one or two carotid arteries

Exclusion Criteria:

* Planned associated valve surgery or concurrent carotid endarterectomy
* Planned aortic dissection repair or aortic root reconstruction
* Screening visit occurring less than 4 hours before scheduled CABG surgery
* MMSE score less than 24 at the screening visit
* Current cardiogenic shock, acute left ventricular rupture, ventricular septal rupture, or papillary muscle rupture
* Uncontrolled diabetes defined as fasting serum blood glucose value equal to or greater than 24 mmol/L (432 mg/dL) at the time of screening (if fasting serum blood glucose not obtained at screening, values obtained within 30 days prior to screening visit may be used)
* Myocardial infarction occurring <48 hours prior to planned CABG surgery
* Severe renal dysfunction defined as a serum creatinine value ≥ 250 micromol/L (2.8 mg/dL) or nephritic syndrome at screening (or obtained within 30 days prior to screening visit)
* History of liver cirrhosis, chronic active hepatitis, or severe liver dysfunction , or liver transaminase ≥3 times ULN at screening (or obtained within 30 days prior to screening visit)
* History of malignancy during last 5 years except for basal cell carcinoma
* Planned surgery for atrial fibrillation
* Pregnancy or potential for pregnancy
* Any medical or psychiatric condition which in the opinion of the investigator makes the patient an unsuitable candidate for the study
* History of alcohol or drug abuse within the past year
* Participation in any other investigation drug or device study within 30 days of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2004-04; Study Completion 2005-10

PRIMARY OUTCOMES:
Combined incidence of cardiovascular death, nonfatal myocardial infarction and nonfatal cerebral infarction on days up to and including post-operative day 30.

SECONDARY OUTCOMES:
Combined incidence of cardiovascular death, nonfatal myocardial infarction and nonfatal cerebral infarction up to and including post-operative day (POD) 90
Incidence of cardiovascular death up to and including POD 4, POD 30, POD 90
Incidence of nonfatal myocardial infarction up to and including POD 4, POD 30, POD 90
Incidence of all cause morality up to and including POD 4, POD 30, POD 90
Global disability as measured by the Modified Rankin scale at POD 30 and POD 90
MMSE score at POD 30 and POD 90
Among patients with a confirmed cerebral infarction, severity of stroke as measured by the National Institutes of Health Stroke Scale (NIHSS) at the time of stroke diagnosis and at subsequent study visits up to and including POD 90
Psychometric testing results as measured by a short battery of tests at POD 4, POD 30 and POD 90 on a subset of approximately 150 volunteers per treatment arm
CK-MB AUC (0-24 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD, FRCPC, FACC, Principal Investigator — Montreal Heart Institute Research Centre
Locations (2):
- Duke University Medical Center, Durham, North Carolina, United States
- Montreal Heart Institute, Montreal, Quebec, Canada